CLINICAL TRIAL: NCT04719936
Title: Comparison Between Superior and Inferior Capsulotomy in Bipolar Hemiarthroplasty Using Posterior Approach
Brief Title: Superior and Inferior Capsulotomy in Bipolar Hemiarthroplasty Using Posterior Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ajou University School of Medicine (Other); Nowon Eulji Medical Center (Unknown); Dankook University (Other); Konkuk University Medical Center (Other); Gyeongsang National University Hospital (Other); Semyeong Christianity Hospital (Unknown)
Responsible Party: Principal Investigator, Young-Kyun Lee, Professor, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAICO study
Record Dates: First submitted 2021-01-12; First posted 2021-01-22 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2023-04

CONDITIONS: Femoral Neck Fractures
Keywords: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Intervention Model Description: Inferior capsulotomy in bipolar hemiarthroplasty will be performed in 25 patients.
  As control group, historical group of patients who received bipolar hemiarthroplasty using superior capsulotomy from January 2010 to December 2020 will be included. A total of 5500 patients are to be included in multicenters.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- inferior capsulotomy group (Experimental): inferior capsulotomy will be conducted during posterior approach.
  Interventions: Procedure: inferior capsulotomy
- superior capsulotomy group (Active Comparator): superior capsulotomy was conducted during posterior approach. (These control group is consisted of patients who received bipolar hemiarthroplasty using superior capsulotomy from January 2010 to December 2020)
  Interventions: Procedure: superior capsulotomy

INTERVENTIONS:
Procedure: inferior capsulotomy — inferior capsulotomy will be conducted during posterior approach.
  Arms: inferior capsulotomy group
Procedure: superior capsulotomy — superior capsulotomy was conducted during posterior approach. (These control group is consisted of patients who received bipolar hemiarthroplasty using superior capsulotomy from January 2010 to December 2020)
  Arms: superior capsulotomy group

SUMMARY:
Investigators will compared the clinical outcomes between superior capulotomy and inferior capsulotomy in bipolar hemiarthropalsty using posterior approach.

DETAILED DESCRIPTION:
primary clinical outcome will be dislocation within 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* more than 50 years old
* displaced femoral neck fractgure

Exclusion Criteria:

* less than 50 years old

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3502 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
dislocation | 12 months
  rate of dislocation

SECONDARY OUTCOMES:
mobility change | 12 months
  change of mobility according to Koval classification; independent community ambulatory community ambulatory with cane community ambulatory with crutch, walker independent household ambulatory household ambulatory with cane household ambulatory with crutch, walker nonfunctional ambulatory

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No